CLINICAL TRIAL: NCT07048847
Title: The Effect of Supervised Aerobic Exercise on Adipokine and Myokine Biomarkers in Patients With Cancer During Systemic Chemotherapy
Brief Title: The Effect of Aerobic Exercise on Selective Biomarkers of Patients With Cancer
Status: Completed | Type: Observational
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Alper Tuğral, Project Coordinator, Izmir Bakircay University
Other Study IDs: BakircayU-579/559
Record Dates: First submitted 2025-06-10; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Colon Cancer; Chemotherapy Effect
Keywords: Adiponectin; Cancer; Exercise; Irisin; IL-6; Leptin
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — For both EG and CG, two blood samplings were performed for each patient. 5 cc venous blood was collected from all the participants and centrifuged at 1500 g for 10 minutes. Separated serum was stored at -20 °C until analysis. Serum leptin, IL-6, irisin, and adiponectin concentrations were measured by using enzyme-linked immunosorbent assay (ELISA) method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exercise Group: Patients who will be willing to participate in supervised exercise will be grouped in Exercise Group (EG).
  Interventions: Other: Exercise
- Control Group: Patients who are not willing to participate in exercise due to various reasons (time restrictions, other obligations, transport, etc.) will be grouped in the Control Group (CG).

INTERVENTIONS:
Other: Exercise — The exercise program will be started with 25 Watt (W) for 5 minutes of warm-up. Then it is steadily increased automatically by 5W in 5 minutes apart for 25 minutes for the loading period. The last 5 minutes which will be started by lowering the load to 25 W for cooling will be implemented for cooling down. To prevent acommodation, the warm-up period will be modified by increasing nearly 10% of its previous rate three weeks apart.A submaximal exercise prescription will be followed according to the American College of Sports Medicine guideline by taking into attention 50-70% of Heart Rate Reserve.A submaximal exercise prescription will be followed according to the American College of Sports Medicine guideline by taking into attention 50-70% of Heart Rate Reserve.
  Other Names: Control
  Groups: Exercise Group

SUMMARY:
This study is a single-blinded, prospective, controlled trial aiming to evaluate the effect of supervised aerobic exercise on adipokine and myokine biomarkers in patients with breast or colon cancer during their systemic chemotherapy.

DETAILED DESCRIPTION:
To determine the effect of aerobic exercise on adipokine and myokine biomarkers such as Interleukin-6 (IL-6), Irisin, Leptin and Adiponectin in the blood of breast or colon cancer patients receiving chemotherapy compared to ones who did not exercise during their systemic chemotherapy.

Patients who were diagnosed with solid type of cancer specifically focusing on breast or colon cancer will be recruited either to the exercise group (EG) or control group (CG) during their systemic chemotherapy. An individualized supervised resistive aerobic exercise which will be performed via stationary resistive biycle ergometer will be implemented along with the chemotherapy process for EG.

Each exercise session will be performed 2 times per week for at least 12 weeks (can be extended up to 24 weeks) during chemotherapy.

Exercise intensity will be set as submaximal, 50-70% of heart rate reserve, and each session will be lasted 35 minutes.

All exercise sessions will be supervised by the researchers to avoid potential side effects.

5 cc venous blood samples will be collected before the first and last chemotherapy infusions (for both EG and CG). The samples will be blinded to the analyzers did not know which group the samples belonged to.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with solid type of cancer
* Being candidate for systemic chemotherapy
* Being volunteer to participate in an exercise program
* Aged between 18-70 years old

Exclusion Criteria:

* Having 2 or above grades according to the Eastern Cooperative Oncology Group (ECOG) performance status
* Having mental and/or cognitive deficits
* Ongoing medical and/or surgical (if any) complications
* Having neurological/orthopedical and/or severe respiratory dysfunctions
* Having any condition which corresponds to the contraindication of exercise (i.e. advanced stages, distant metastasis, infection)
* Having unstable vital parameters or having regularly used pharmacological interventions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Having been diagnosed with solid type of cancer (specifically breast or colon) and being candidate for undergoing systemic chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Irisin | Baseline
  Measuring Serum levels of Irisin via ELISA
Irisin | From completion of systemic chemotherapy up to one week
  Measuring Serum levels of Irisin via ELISA
Leptin | Baseline
  Measuring Serum levels of Leptin via ELISA
Leptin | From completion of systemic chemotherapy up to one week
  Measuring Serum levels of Leptin via ELISA
Adiponectin | Baseline
  Measuring Serum levels of Adiponectin via ELISA
Adiponectin | From completion of systemic chemotherapy up to one week
  Measuring Serum levels of Adiponectin via ELISA
Interleukin-6 (IL-6) | Baseline
  Measuring Serum levels of IL-6 via ELISA
Interleukin-6 (IL-6) | From completion of systemic chemotherapy up to one week
  Measuring Serum levels of IL-6 via ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Alper Tuğral, PhD, Principal Investigator — Izmir Bakircay University
Locations (1):
- Bakircay University Çiğli State and Training Hospital, Department of Medical Oncology, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The data can be available with a reasonable request as well as the permission of the ethical board

REFERENCES:
- [Background] Brownson-Smith R, Orange ST, Cresti N, Hunt K, Saxton J, Temesi J. Effect of exercise before and/or during taxane-containing chemotherapy treatment on chemotherapy-induced peripheral neuropathy symptoms in women with breast cancer: systematic review and meta-analysis. J Cancer Surviv. 2025 Feb;19(1):78-96. doi: 10.1007/s11764-023-01450-w. Epub 2023 Aug 24. PMID 37615928
- [Background] Kim JS, Galvao DA, Newton RU, Gray E, Taaffe DR. Exercise-induced myokines and their effect on prostate cancer. Nat Rev Urol. 2021 Sep;18(9):519-542. doi: 10.1038/s41585-021-00476-y. Epub 2021 Jun 22. PMID 34158658
- [Background] Tsiani E, Tsakiridis N, Kouvelioti R, Jaglanian A, Klentrou P. Current Evidence of the Role of the Myokine Irisin in Cancer. Cancers (Basel). 2021 May 27;13(11):2628. doi: 10.3390/cancers13112628. PMID 34071869
- [Background] Dieli-Conwright CM, Courneya KS, Demark-Wahnefried W, Sami N, Lee K, Buchanan TA, Spicer DV, Tripathy D, Bernstein L, Mortimer JE. Effects of Aerobic and Resistance Exercise on Metabolic Syndrome, Sarcopenic Obesity, and Circulating Biomarkers in Overweight or Obese Survivors of Breast Cancer: A Randomized Controlled Trial. J Clin Oncol. 2018 Mar 20;36(9):875-883. doi: 10.1200/JCO.2017.75.7526. Epub 2018 Jan 22. PMID 29356607
- [Background] Meneses-Echavez JF, Correa-Bautista JE, Gonzalez-Jimenez E, Schmidt Rio-Valle J, Elkins MR, Lobelo F, Ramirez-Velez R. The Effect of Exercise Training on Mediators of Inflammation in Breast Cancer Survivors: A Systematic Review with Meta-analysis. Cancer Epidemiol Biomarkers Prev. 2016 Jul;25(7):1009-17. doi: 10.1158/1055-9965.EPI-15-1061. Epub 2016 Apr 12. PMID 27197276
- [Background] Tjoe JA, Piacentine LB, Papanek PE, Raff H, Richards J, Harkins AL, Yin J, Ng AV. Team triathlon effects on physiological, psychological, and immunological measures in women breast cancer survivors. Support Care Cancer. 2020 Dec;28(12):6095-6104. doi: 10.1007/s00520-020-05457-2. Epub 2020 Apr 20. PMID 32314053
- [Derived] Tugral A, Aribas Z, Kaya Ucar G, Arslan FD, Bakar Y, Karakoyun I, Akyol M. The effect of supervised aerobic exercise on adipokine and myokine biomarkers in patients with cancer during systemic chemotherapy: a single-blinded prospective controlled trial. Support Care Cancer. 2025 Aug 2;33(8):741. doi: 10.1007/s00520-025-09788-w. PMID 40751845